CLINICAL TRIAL: NCT00093509
Title: Magnetic Resonance Based Non-Invasive Thermometry for Hyperthermic Treatment of Extremity Soft Tissue Sarcomas: A Multimodal Phase I/II Study
Brief Title: MRI Sarcoma Non Invasive Thermometry
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mark Dewhirst (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mark Dewhirst, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008831; DUMC-1308-04-7R5 (Other: Legacy Duke IRB number from paper system); DUMC-G880018; CDR0000388048 (Other: National Cancer Institute (NCI))
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Sarcoma
Keywords: stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide; Mesna; Diathermy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic Resonance Based Thermometry (Experimental): Patients will receive hyperthermia throughout the course of radiotherapy delivered once weekly for a total of 5 treatments. Each treatment will last 1-2 hours with a goal of delivering a cumulative thermal dose of 10-100 CEM 43˚T90. Interstitial temperature measurements will be taken by placing a single (less than or equal to) 15 gauge thermometry catheter into the tumor.
  In addition to hyperthermia treatment and radiation therapy all patients will receive conventional surgery for the removal of their tumors. Some patients will also receive chemotherapy if their treating physician thinks it is the their best interested (including the possibility of doxorubicin hydrochloride or ifosfamide and mesna).
  Interventions: Drug: doxorubicin hydrochloride; Drug: ifosfamide and mesna; Procedure: hyperthermia treatment with an MRI Compatible Radiofrequency Extremity Hyperthermia Applicator; Radiation: radiation therapy

INTERVENTIONS:
Drug: doxorubicin hydrochloride — To be dosed at 75 mg/m2 i.v. push every 4 weeks for 4 cycles. This treatment is optional and will not be used on all subjects.
  Other Names: Adriamycin
Drug: ifosfamide and mesna — 2 gm / m2 ifosfamide mixed in 1000 cc D5W infused continuously over 24 hours daily for 6 days (144 hours); total ifosfamide dose 12 gm/ m2. For the day infusion only MESNA (sodium 2-mercapto-ethanesulphonate) is mixed with ifosfamide as above and given at 2.5 gm / m2 / 24 hours.
  Other Names: Ifosfamide - Ifex; Mesna - sodium 2-mercapto-ethanesulphonate
Procedure: hyperthermia treatment with an MRI Compatible Radiofrequency Extremity Hyperthermia Applicator — Patients will receive hyperthermia throughout the course of radiotherapy delivered once weekly for a total of 5 treatments. Each treatment will last 1-2 hours with a goal of delivering a cumulative thermal dose of 10-100 CEM 43˚T90.
Radiation: radiation therapy — External beam megavoltage (≥ 4 MV) beams will be used at SSD, SAD ≥ 70 cm at a dose rate of > 100 cGy/min. Fraction sizes of 180 cGy will be used 5 times per weeks in a continuous course. Total dose will be 45 Gy + 10%, consistent with sites being treated.

SUMMARY:
RATIONALE: Hyperthermia therapy kills tumor cells by heating them to several degrees above body temperature. Using MRI to measure heat may help to determine the effectiveness of hyperthermia therapy. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as ifosfamide and doxorubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining hyperthermia with radiation therapy and chemotherapy before surgery may kill more tumor cells and shrink the tumor so that it can be removed.

PURPOSE: This phase I/II trial is studying the side effects of hyperthermia when given together with radiation therapy and optional chemotherapy and to see how well they work in treating patients who are undergoing surgery for soft tissue sarcoma of the limbs.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and accuracy of real time magnetic resonance-based non-invasive thermometry in patients with grade 2 or 3 soft tissue sarcoma of the extremity receiving combination hyperthermia, radiotherapy, surgery, and optional high-dose ifosfamide and doxorubicin.

Secondary

* Determine the local control, disease-free survival, and overall survival of patients treated with this regimen.
* Determine acute and late toxic effects of this regimen in these patients.
* Correlate measurements of tumor physiology, defined by gadolinium-enhanced magnetic resonance imaging, magnetic resonance spectroscopy, and tumor oxygenation, with clinical and/or pathological response and/or metastatic potential in patients treated with this regimen.

OUTLINE: Patients may receive high-dose ifosfamide IV continuously over 6 days (144 hours). Beginning 3 weeks after the completion of ifosfamide, patients undergo radiotherapy once daily, 5 days a week, for 5 weeks. Beginning 1 hour after radiotherapy, patients also undergo hyperthermia (with heat measured by conventional and magnetic resonance-based thermometry) over 1-2 hours once weekly for 5 weeks. Approximately 4 weeks after the completion of radiotherapy and hyperthermia, patients undergo surgery. Approximately 1 month after surgery, patients may then receive high-dose doxorubicin IV once every 4 weeks for 4 courses.

PROJECTED ACCRUAL: A total of 10-30 patients will be accrued for this study within 2-6 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have histologically proven grade 2 or grade 3 soft tissue sarcoma.
* Karnofsky performance status ≥ 70.
* Life expectancy ≥ 6 months.
* There is no specific tumor size limitation, but the involved extremity must fit within the hyperthermia applicator.
* Patients must be ≥ 18 years of age.
* Patients who are to receive chemotherapy must have a left ventricular ejection fraction on resting MUGA scan of at least 45% to confirm adequate cardiac function
* Patients must competent to consent to be in the study and sign an approved informed consent.

Exclusion Criteria:

* Pregnant patients
* Patients with cardiac pacemakers and implanted defibrillators or other devices not compatible with ultrasound or microwave technology
* Patients who have any metal in their bodies including orthopedic rods, surgical clips, bullets, or shrapnel, etc. unless cleared by MRI staff and Hyperthermia physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1999-11; Primary Completion 2007-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Temperature Rise from Baseline | 1 hour
  MR-based thermometry measures: We are assessing agreement between the non-invasive MR measurements versus the invasive interstitial point measurements. The equivalence of median temperature measured within one or more MR ROI's (regions-of-interest in the MR image) and temperatures measured invasively in tissue immediately adjacent to those ROI's;

SECONDARY OUTCOMES:
Overall Survival | every 6 months for up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ellen L. Jones, MD, PhD, Principal Investigator — Duke Cancer Institute; Zeljko Vujaskovic, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

REFERENCES:
- [Result] Craciunescu OI, Stauffer PR, Soher BJ, Wyatt CR, Arabe O, Maccarini P, Das SK, Cheng KS, Wong TZ, Jones EL, Dewhirst MW, Vujaskovic Z, MacFall JR. Accuracy of real time noninvasive temperature measurements using magnetic resonance thermal imaging in patients treated for high grade extremity soft tissue sarcomas. Med Phys. 2009 Nov;36(11):4848-58. doi: 10.1118/1.3227506. PMID 19994492